CLINICAL TRIAL: NCT00884741
Title: Phase III Double-blind Placebo-Controlled Trial of Conventional Concurrent Chemoradiation and Adjuvant Temozolomide Plus Bevacizumab Versus Conventional Concurrent Chemoradiation and Adjuvant Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Temozolomide and Radiation Therapy With or Without Bevacizumab in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-01670; NCI-2009-01670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-0825; RTOG 0825; CDR0000640428; RTOG-0825 (Other: NRG Oncology); RTOG-0825 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Glioblastoma; Gliosarcoma; Supratentorial Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; Bevacizumab; Immunoglobulin G; Disulfides; Radiotherapy, Intensity-Modulated; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (radiation therapy, temozolomide, placebo) (Active Comparator): Patients undergo intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy 5 days a week for 6 weeks and receive temozolomide PO QD for up to 7 weeks. Beginning 4 weeks after completion of chemotherapy and radiation therapy, patients receive temozolomide PO QD on days 1-5. Treatment with temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive placebo IV over 30-90 minutes once every 2 weeks beginning in week 4 of chemotherapy and radiation therapy and continuing until the completion of temozolomide.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Quality-of-Life Assessment; Drug: Temozolomide
- Arm II (radiation therapy, temozolomide, bevacizumab) (Experimental): Patients undergo radiation therapy and receive temozolomide as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning in week 4 of chemoradiotherapy and continuing until the completion of adjuvant temozolomide.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Biological: Bevacizumab; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Temozolomide

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3-dimentional conformal radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm II (radiation therapy, temozolomide, bevacizumab)
Radiation: Intensity-Modulated Radiation Therapy — Undergo intensity-modulated radiation therapy
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I (radiation therapy, temozolomide, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Temozolomide — Given orally
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This randomized phase III trial studies temozolomide (TMZ) and radiation therapy (RT) to compare how well they work with or without bevacizumab in treating patients with newly diagnosed glioblastoma or gliosarcoma. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as bevacizumab, may find tumor cells and help kill them. It is not yet known whether temozolomide and radiation therapy are more effective when given together with or without bevacizumab in treating glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of bevacizumab to temozolomide and radiation improves efficacy as measured by progression-free and/or overall survival.

II. To assess the association between overall survival and K^trans change from T1 to T2. (ACRIN 6686) III. To assess the association between overall survival and spin echo cerebral blood volume (CBV) change from T1 to T2. (ACRIN 6686)

SECONDARY OBJECTIVES:

I. To determine whether the tumor molecular profile conferring a mesenchymal/angiogenic phenotype is associated with a selective increase in benefit, as measured by either overall survival or progression-free survival, from the addition of bevacizumab.

II. To compare and record the toxicities of the conventional and bevacizumab-containing regimens.

III. To assess the association between progression-free survival and K^trans change from T1 to T2. (ACRIN 6686) IV. To assess the association between progression-free survival and spin echo CBV change from T1 to T2. (ACRIN 6686) V. To assess the association between values of K^trans and spin echo CBV measured separately at T0 and at T1, and overall and progression-free survival. (ACRIN 6686) VI. To assess the association between overall survival and K^trans changes from T0 to T1 and from T2 to T3. (ACRIN 6686) VII. To assess the association between overall survival and spin echo CBV changes from T0 to T1 and from T2 to T3. (ACRIN 6686) VIII. To assess the association between overall survival and apparent diffusion coefficient (ADC) change from T0 to T1. (ACRIN 6686) IX. To assess the association between overall survival and ADC change from T1 to T2. (ACRIN 6686) X. To assess the association between progression-free survival and ADC change from T0 to T1. (ACRIN 6686) XI. To assess the association between progression-free survival and ADC change from T1 to T2. (ACRIN 6686) XII. To assess the association between T1 values of ADC and overall and progression-free survival. (ACRIN 6686) XIII. To assess the association between change in lesion size between T1 and T3, as measured by advanced magnetic resonance imaging (MRI), and overall and progression-free survival. (ACRIN 6686)

TERTIARY OBJECTIVES:

I. To determine the differential acute effects associated with the addition of bevacizumab to temozolomide and radiation, as compared to the conventional arm, on measures of neurocognitive function, health-related quality of life, and symptoms during radiation and across the longitudinal progression-free interval.

II. To determine the relationship of neurocognitive function, health-related quality of life, and symptoms, with progression-free and overall survival.

III. To determine the association between tumor molecular profile (i.e., mesenchymal/angiogenic phenotype and proneural phenotype) and neurocognitive function, health-related quality of life, and symptoms.

IV. To describe the association between health-related quality of life as measured by the European Organization for Research and Treatment Quality of Life Questionnaire-Core 30/Brain Cancer Module-20 (EORTC-QL30/BCM20) and mean symptom severity as measured by the M. D. Anderson Symptom Inventory Brain Tumor Module (MDASI-BT) in patients enrolled in this study.

V. To evaluate the relationship between self-reported neurocognitive function and objectively measured tests of neurocognitive function (NCF).

VI. To assess the association between measures of change in enhancing tumor size at week 22 and overall survival in participants with glioma receiving chemoradiotherapy with and without bevacizumab.

VII. To assess the association between measures of change in T2-based tumor size at week 22 and overall survival in participants with glioma receiving chemoradiotherapy with and without bevacizumab.

VIII. To assess the association between changes in ADC values and overall survival in participants with glioma receiving chemoradiotherapy with and without bevacizumab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms (there are also two registration steps prior to randomization which are labeled as "arms" in ClinicalTrials.gov to facilitate entry of results into the website).

ARM I: Patients undergo intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy 5 days a week for 6 weeks and receive temozolomide orally (PO) once daily (QD) for up to 7 weeks. Beginning 4 weeks after completion of chemotherapy and radiation therapy, patients receive temozolomide PO QD on days 1-5. Treatment with temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive placebo IV over 30-90 minutes once every 2 weeks beginning in week 4 of chemotherapy and radiation therapy and continuing until the completion of temozolomide.

ARM II: Patients undergo radiation therapy and receive temozolomide as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning in week 4 of chemoradiotherapy and continuing until the completion of adjuvant temozolomide.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of glioblastoma or gliosarcoma (World Health Organization [WHO] grade IV) confirmed by central review prior to step 2 registration
* Tumor tissue that is determined by central pathology review prior to step 2 registration to be of sufficient size for analysis of O-6-methylguanine-DNA methyltransferase (MGMT) and determination of molecular profile

  * Patients must have at least 1 block of tumor tissue; submission of 2 blocks is strongly encouraged to maximize the chances of eligibility; at least 1 cubic centimeter of tissue composed primarily of tumor must be present
  * CUSA (Cavitron ultrasonic aspirator)-derived material is not allowed; fresh frozen tumor tissue acquisition is encouraged
  * Diagnosis must be made by surgical excision, either partial or complete; stereotactic biopsy is not allowed because it will not provide sufficient tissue for MGMT analysis
  * The tumor tissue should be sent as soon as possible to maximize the likelihood of eligibility; tumor tissue should be submitted by 4 weeks after the surgical procedure so that the study registration and treatment can commence by the mandatory 5 week post-surgery outer limit
  * Sites must submit tissue fir central review in order to obtain the MGMT analysis; patients from sites not following protocol-specified process for obtaining MGMT results will be made ineligible
* The tumor must have a supratentorial component
* History/physical examination within 14 days prior to step 2 registration
* The patient must have recovered from the effects of surgery, postoperative infection, and other complications before step 2 registration
* A diagnostic contrast-enhanced MRI of the brain must be performed preoperatively and postoperatively prior to the initiation of radiotherapy; the postoperative scan must be performed within 28 days prior to step 1 registration

  * An MRI or computed tomography (CT) scan (potentially in addition to the postoperative scan) must be obtained within 10 days prior to the start of radiation therapy and must not demonstrate significant postoperative hemorrhage defined as > 1 cm diameter of blood; if > 1 cm of acute blood is detected, the patient will be ineligible for this trial; the radiation planning MRI or CT scan may be used to determine presence of hemorrhage
  * Patients unable to undergo MR imaging because of non-compatible devices can be enrolled, provided pre- and postoperative contrast-enhanced CT scans are obtained and are of sufficient quality; preoperative and postoperative scans must be the same type; such patients cannot be enrolled into the advanced imaging component
* Documentation of steroid doses within 14 days prior to step 2 registration
* Karnofsky performance status >= 70
* Absolute neutrophil count (ANC) >= 1,800 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 10.0 g/dL (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable)
* Blood urea nitrogen (BUN) =< 30 mg/dL within 14 days prior to step 2 registration
* Creatinine =< 1.7 mg/dl within 14 days prior to step 2 registration
* Urine protein screened by urine analysis for urine protein creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg
* Bilirubin =< 2.0 mg/dl within 14 days prior to step 2 registration
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 3 x normal range within 14 days prior to step 2 registration
* Systolic blood pressure =< 160 mg Hg or diastolic pressure =< 90 mm Hg within 14 days prior to step 2 registration
* Electrocardiogram without evidence of acute cardiac ischemia within 14 days prior to step 2 registration
* Prothrombin time/international normalized ratio (PT INR) < 1.4 for patients not on warfarin confirmed by testing within 14 days prior to step 2 registration
* Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight [LMW] heparin) must meet both of the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * In-range INR (between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of LMW heparin
* Patient must provide study specific informed consent prior to study entry
* Women of childbearing potential and male participants must practice adequate contraception
* For females of child-bearing potential, negative serum pregnancy test within 14 days prior to step 2 registration

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for >= 3 years; (for example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible)
* Recurrent or multifocal malignant gliomas
* Metastases detected below the tentorium or beyond the cranial vault
* Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable, except prior temozolomide or bevacizumab; prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted
* Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 14 days of step 2 registration
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to step 2 registration
  * History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy
  * Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to step 2 registration, with the exception of the craniotomy for tumor resection
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of step 2 registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * Acquired immune deficiency syndrome (AIDS) based upon current Center for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive
  * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
  * Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Pregnant or lactating women
* Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study
* For American College of Radiology Imaging Network (ACRIN) 6686 Advanced Imaging: inability to undergo MRI (e.g., due to safety reasons, such as presence of a pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2013-03-17 (Actual); Study Completion 2013-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gilbert, Principal Investigator — NRG Oncology
Locations (330):
- United States (324):
  - Providence Hospital, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center - North Fresno, Fresno, California
  - Cancer Care Associates of Fresno Medical Group Inc, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Cape Radiation Oncology, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Concord Hospital, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - South Nassau Communities, Oceanside, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Highland Hospital, Rochester, New York
  - University Radiation Oncology, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - University Pointe, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Texas Oncology Methodist Charlton Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - West Texas Cancer Center, Odessa, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Radiology Associates of Appleton/ThedaCare Regional Medical Center, Appleton, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
- Canada (5):
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Health Sciences North, Greater Sudbury, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317

RESULTS

PARTICIPANT FLOW:
Groups:
- Step 1 Registration: No treatment. Central Pathology Tissue Screening to confirm histology and adequacy of tissue for MGMT analysis and molecular profile. Tumor tissue must be received and central review confirmation completed before STEP 2 registration can occur.
- Step 2 Registration: Pre-Randomization TMZ+RT: Temozolomide pre-randomization, radiation therapy pre-randomization
- Randomized Arm 1: TMZ+RT + Placebo: Temozolomide post-randomization,Radiation therapy post-randomization, placebo
- Randomized Arm 2: TMZ+RT + Bevacizumab: Temozolomide post-randomization, radiation therapy post-randomization, bevacizumab
Period: Step 1 Registration: Tissue Screening
Arm/Group | Step 1 Registration | Step 2 Registration: Pre-Randomization TMZ+RT | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Started | 978 | 0 | 0 | 0
Completed | 666 | 0 | 0 | 0
Not Completed | 312 | 0 | 0 | 0
Not completed — Protocol Violation | 157 | 0 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0
Not completed — Insufficient tissue | 105 | 0 | 0 | 0
Not completed — Disease progression | 12 | 0 | 0 | 0
Not completed — Patient refusal | 32 | 0 | 0 | 0
Period: Step 2 Registration: Tissue Analysis
Arm/Group | Step 1 Registration | Step 2 Registration: Pre-Randomization TMZ+RT | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Started | 0 (Step 1 Registration Arm goes to Step 2 Registration Arm) | 666 (These patients completed the previous period on the Step 1 Registration arm.) | 0 | 0
Completed | 0 | 637 | 0 | 0
Not Completed | 0 | 29 | 0 | 0
Not completed — Protocol Violation | 0 | 15 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Patient refusal | 0 | 7 | 0 | 0
Not completed — Disease Progression | 0 | 4 | 0 | 0
Period: Randomization
Arm/Group | Step 1 Registration | Step 2 Registration: Pre-Randomization TMZ+RT | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Started | 0 | 0 (Step 2 Registration Arm goes to a randomized arm.) | 317 (These patients completed the previous period on the Step 2 Registration arm.) | 320 (These patients completed the previous period on the Step 2 Registration arm.)
Completed | 0 | 0 | 309 (Patients with data available for the primary analysis are considered to have completed the study.) | 312 (Patients with data available for the primary analysis are considered to have completed the study.)
Not Completed | 0 | 0 | 8 | 8
Not completed — Protocol Violation | 0 | 0 | 8 | 8

BASELINE CHARACTERISTICS:
Population: All eligible patients. Note that the Pre-Randomization TMZ+RT arm only includes eligible patients that did not continue to randomization.
Groups:
- Pre-Randomization TMZ+RT: Temozolomide pre-randomization, radiation therapy pre-randomization. Note that for the purpose of this table, this arm only includes patients that did not continue to randomization.
- Total: Total of all reporting groups
Arm/Group | Pre-Randomization TMZ+RT | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab | Total
Number analyzed (Participants) | 29 | 309 | 312 | 650
Age, Continuous [Median (Full Range); unit: years] | 58 [25 to 75] | 57 [19 to 82] | 59 [21 to 82] | 58 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 115 | 134 | 260
  Male | 18 | 194 | 178 | 390

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Survival time was defined as time from randomization to date of death from any cause and was estimated by the Kaplan-Meier method. Patients last known to be alive were censored at the date of last contact. This analysis was planned to occur when 390 deaths had been reported.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs after all 390 deaths have been reported.
Population: All eligible randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Number analyzed (Participants) | 309 | 312
months | 16.1 [14.8 to 18.7] | 15.7 [14.2 to 16.8]
Statistical Analysis 1: Comparison: Randomized Arm 1: TMZ+RT + Placebo vs Randomized Arm 2: TMZ+RT + Bevacizumab; The trial was designed to concurrently provide 80% power for the detection of a 25% relative reduction in mortality hazard (hazard ratio .75) and 30% reduction in progression hazard (hazard ratio .70) for the addition of bevacizumab to temozolomide and radiation. To control for type I error in testing the co-primary endpoints, the significance criterion for OS was 0.023 (one-sided) and for PFS was 0.002 (one-sided); Test type: Superiority or Other; p = 0.11, Log Rank — To control for type I error in testing the co-primary endpoints, the significance criterion for OS was 0.023 (one-sided) and for PFS was 0.002 (one-sided); Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.93 to 1.37]

2. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as time from randomization to date of progression, death, or last follow-up, and was estimated by the Kaplan-Meier method. Patients last known to be alive were censored at the date of last contact. This analysis was planned to occur when 390 deaths had been reported.
Time Frame: From randomization to date of progression, death, or last follow-up for progression-free survival. Analysis occurs after all 390 deaths have been reported.
Population: All eligible randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Number analyzed (Participants) | 309 | 312
months | 7.3 [5.6 to 7.9] | 10.7 [10.0 to 12.2]
Statistical Analysis 1: Comparison: Randomized Arm 1: TMZ+RT + Placebo vs Randomized Arm 2: TMZ+RT + Bevacizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.79, 95% CI 2-sided [0.66 to 0.94]

3. Secondary Outcome: Incidence of Grade 3 and Higher Treatment-related Toxicity as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (AEs) Version 3.0
Description: AEs are graded by using CTCAE 3.0. The difference between the two randomized arms in the percentage of patients with grade 3 or higher toxicities reported as possibly/probably/definitely related to protocol treatment will be tested using a chi square test.
Time Frame: Up to 30 days
Population: Eligible randomized patients with adverse event data who started study treatment.
Measure: Number; unit: participants
Arm/Group | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Number analyzed (Participants) | 300 | 303
participants | 87 | 97
Statistical Analysis 1: Comparison: Randomized Arm 1: TMZ+RT + Placebo vs Randomized Arm 2: TMZ+RT + Bevacizumab; Test type: Superiority or Other; p = 0.42, Chi-squared — Two-sided

4. Other Pre Specified Outcome: Quality of Life Measured by the M.D. Anderson Symptom Inventory Brain Tumor Module (MDASI-BT Tool) and EORTC Quality of Life Questionnaire-Core/Brain Cancer Module( QLQ-C30/BCM20)
Time Frame: Analysis can occur at or after time of primary outcome measure analysis.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Neurocognitive Function Measured by the Hopkins Verbal Learning Test-Revised(HVLT-R), Trail Making Test Part A, Trail Making Test Part B, Controlled Oral Word Association Test (COWAT)
Time Frame: Analysis can occur at or after time of primary outcome measure analysis.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Data is reported for eligible randomized patients with adverse event data who started study treatment. Subjects experiencing more than one of a given serious adverse event (SAE) were counted only once for that SAE. The same methodology was applied for non-serious adverse events.
Arm/Group | Pre-Randomization TMZ+RT | Randomized Arm 1: TMZ+RT + Placebo | Randomized Arm 2: TMZ+RT + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 5/10 | 115/300 | 141/303
Other Adverse Events (participants affected / at risk) | 7/10 | 292/300 | 292/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Randomization TMZ+RT (N=10) | Randomized Arm 1: TMZ+RT + Placebo (N=300) | Randomized Arm 2: TMZ+RT + Bevacizumab (N=303)
Blood disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 2 | 9
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 8
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Myocardial ischemia (Cardiac disorders) | 0 | 2 | 2
Dry eye syndrome (Eye disorders) | 0 | 1 | 0
Eye disorder (Eye disorders) | 1 | 2 | 0
Retinal detachment (Eye disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 4
Cecal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1 | 5
Constipation (Gastrointestinal disorders) | 0 | 7 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 10
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 6
Chest pain (General disorders) | 0 | 1 | 2
Death (General disorders) | 0 | 2 | 8
Disease progression (General disorders) | 1 | 5 | 2
Edema limbs (General disorders) | 0 | 1 | 2
Fatigue (General disorders) | 0 | 15 | 16
Fever (General disorders) | 0 | 5 | 4
Gait abnormal (General disorders) | 0 | 2 | 2
Localized edema [head and neck] (General disorders) | 0 | 1 | 0
Pain [other] (General disorders) | 0 | 1 | 1
Sudden death (General disorders) | 0 | 1 | 1
Visceral edema (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder pain (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 2
Abdominal infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 0
Appendicitis [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Bladder infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Bone infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Catheter related infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Encephalitis infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 1
Eye infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 1
Ileal infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Infection [neck, with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1
Infection [other] (Infections and infestations) | 0 | 2 | 0
Infectious colitis [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1
Infective myositis [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Mucosal infection [with unknown ANC] (Infections and infestations) | 0 | 2 | 0
Opportunistic infection (Infections and infestations) | 0 | 0 | 2
Pancreas infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Peripheral nerve infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Pneumonia [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1
Pneumonia [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Pneumonia [with unknown ANC] (Infections and infestations) | 0 | 3 | 2
Rhinitis infective [with unknown ANC] (Infections and infestations) | 0 | 0 | 1
Sepsis [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1
Sepsis [with unknown ANC] (Infections and infestations) | 0 | 2 | 1
Skin infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 1
Upper aerodigestive tract infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 1
Urinary tract infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1
Urinary tract infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 1
Urinary tract infection [with unknown ANC] (Infections and infestations) | 0 | 1 | 1
Wound infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 2 | 3
Wound infection [with unknown ANC] (Infections and infestations) | 1 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intraoperative hepatobiliary injury - Gallbladder (Injury, poisoning and procedural complications) | 0 | 1 | 0
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 3 | 6
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 4
Cardiac troponin T increased (Investigations) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 2 | 3
Lipase increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 5
Neutrophil count decreased (Investigations) | 0 | 3 | 16
Platelet count decreased (Investigations) | 0 | 1 | 10
Platelet count decreased (Investigations) | 0 | 8 | 29
Weight gain (Investigations) | 0 | 0 | 2
Weight loss (Investigations) | 0 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 7 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 8 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 11
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 4 | 6
Central nervous system necrosis (Nervous system disorders) | 0 | 2 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 4 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 3 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 3
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 3
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 8 | 4
Hydrocephalus (Nervous system disorders) | 0 | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 3 | 4
Ischemia cerebrovascular (Nervous system disorders) | 0 | 4 | 7
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 5 | 2
Mental status changes (Nervous system disorders) | 0 | 1 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Neurological disorder NOS (Nervous system disorders) | 0 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 5 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2
Seizure (Nervous system disorders) | 0 | 23 | 20
Speech disorder (Nervous system disorders) | 0 | 8 | 4
Syncope (Nervous system disorders) | 0 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 10 | 9
Depression (Psychiatric disorders) | 0 | 4 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Psychosis (Psychiatric disorders) | 0 | 0 | 1
Hemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 1
Urogenital disorder (Renal and urinary disorders) | 0 | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 1
Thrombosis (Vascular disorders) | 2 | 22 | 23
Vascular disorder (Vascular disorders) | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Randomization TMZ+RT (N=10) | Randomized Arm 1: TMZ+RT + Placebo (N=300) | Randomized Arm 2: TMZ+RT + Bevacizumab (N=303)
Blood disorder (Blood and lymphatic system disorders) | 0 | 20 | 19
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 | 124 | 111
Leukopenia (Blood and lymphatic system disorders) | 0 | 98 | 119
Lymphopenia (Blood and lymphatic system disorders) | 2 | 96 | 114
Hearing loss (Ear and labyrinth disorders) | 1 | 18 | 20
Tinnitus (Ear and labyrinth disorders) | 1 | 16 | 20
Eye disorder (Eye disorders) | 0 | 25 | 19
Vision blurred (Eye disorders) | 0 | 47 | 47
Abdominal pain (Gastrointestinal disorders) | 0 | 13 | 22
Constipation (Gastrointestinal disorders) | 0 | 126 | 141
Diarrhea (Gastrointestinal disorders) | 0 | 48 | 64
Dry mouth (Gastrointestinal disorders) | 1 | 15 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 21 | 27
Dysphagia (Gastrointestinal disorders) | 1 | 14 | 15
Mucositis oral (Gastrointestinal disorders) | 0 | 15 | 29
Nausea (Gastrointestinal disorders) | 2 | 165 | 184
Vomiting (Gastrointestinal disorders) | 0 | 73 | 82
Chills (General disorders) | 0 | 10 | 24
Edema limbs (General disorders) | 0 | 49 | 43
Fatigue (General disorders) | 3 | 238 | 243
Fever (General disorders) | 0 | 22 | 27
Gait abnormal (General disorders) | 0 | 28 | 22
Localized edema [head and neck] (General disorders) | 0 | 21 | 16
Pain [other] (General disorders) | 0 | 20 | 20
Opportunistic infection (Infections and infestations) | 1 | 2 | 5
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 49 | 42
Fracture (Injury, poisoning and procedural complications) | 1 | 4 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 30 | 47
Alanine aminotransferase increased (Investigations) | 2 | 103 | 93
Alkaline phosphatase increased (Investigations) | 0 | 30 | 30
Aspartate aminotransferase increased (Investigations) | 0 | 69 | 74
CD4 lymphocytes decreased (Investigations) | 0 | 10 | 22
Creatinine increased (Investigations) | 1 | 37 | 35
Hyperbilirubinemia (Investigations) | 0 | 19 | 22
Laboratory test abnormal (Investigations) | 0 | 39 | 39
Neutrophil count decreased (Investigations) | 0 | 19 | 34
Neutrophil count decreased (Investigations) | 0 | 64 | 83
Platelet count decreased (Investigations) | 1 | 47 | 59
Platelet count decreased (Investigations) | 0 | 135 | 171
Weight gain (Investigations) | 0 | 16 | 4
Weight loss (Investigations) | 1 | 39 | 55
Anorexia (Metabolism and nutrition disorders) | 1 | 110 | 127
Dehydration (Metabolism and nutrition disorders) | 0 | 17 | 23
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 114 | 121
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 18 | 24
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 3 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 53 | 53
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 38 | 54
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 14 | 22
Hypokalemia (Metabolism and nutrition disorders) | 0 | 43 | 46
Hyponatremia (Metabolism and nutrition disorders) | 2 | 54 | 73
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 30 | 32
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 33 | 50
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 49 | 58
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 15 | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 26 | 24
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 16 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 18 | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 24 | 44
Acoustic nerve disorder NOS (Nervous system disorders) | 1 | 4 | 0
Ataxia (Nervous system disorders) | 0 | 42 | 45
Cognitive disturbance (Nervous system disorders) | 0 | 25 | 26
Depressed level of consciousness (Nervous system disorders) | 0 | 7 | 23
Dizziness (Nervous system disorders) | 0 | 77 | 75
Headache (Nervous system disorders) | 1 | 155 | 167
Memory impairment (Nervous system disorders) | 1 | 63 | 72
Neurological disorder NOS (Nervous system disorders) | 1 | 25 | 25
Peripheral motor neuropathy (Nervous system disorders) | 0 | 43 | 41
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 50 | 47
Seizure (Nervous system disorders) | 2 | 53 | 61
Speech disorder (Nervous system disorders) | 0 | 56 | 36
Taste alteration (Nervous system disorders) | 1 | 49 | 54
Tremor (Nervous system disorders) | 0 | 31 | 33
Agitation (Psychiatric disorders) | 0 | 27 | 19
Anxiety (Psychiatric disorders) | 0 | 44 | 42
Confusion (Psychiatric disorders) | 0 | 43 | 41
Depression (Psychiatric disorders) | 1 | 36 | 54
Insomnia (Psychiatric disorders) | 0 | 74 | 75
Proteinuria (Renal and urinary disorders) | 0 | 25 | 28
Urinary frequency (Renal and urinary disorders) | 0 | 13 | 24
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 19 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 33 | 50
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 33 | 33
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 15
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 34
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 23
Acne (Skin and subcutaneous tissue disorders) | 0 | 11 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 140 | 169
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 17 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 36 | 35
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 | 36 | 41
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 15 | 13
Hypertension (Vascular disorders) | 1 | 39 | 67
Thrombosis (Vascular disorders) | 2 | 24 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less